CLINICAL TRIAL: NCT00850031
Title: A Prospective, Multicenter Clinical Trial to Evaluate the Safety and Effectiveness of the AcuFocus Corneal Inlay (ACI)™ ACI 7000PDT in Presbyopic Subjects (OUS Study)
Brief Title: Safety and Effectiveness Study of the AcuFocus Corneal Inlay ACI 7000PDT in Presbyopes
Acronym: ACI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AcuFocus, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACU-P08-020A
Record Dates: First submitted 2009-02-20; First posted 2009-02-24 (Estimated); Results first posted 2017-02-06 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-01

CONDITIONS: Presbyopia
Keywords: Presbyopia; Accommodation; Near visual acuity; LASIK
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AcuFocus Corneal Inlay (Experimental): Implantation of the AcuFocus Corneal Inlay in emmetropic presbyopic patients.
  Interventions: Device: AcuFocus Corneal Inlay

INTERVENTIONS:
Device: AcuFocus Corneal Inlay — Inlay implanted in cornea for improvement of near vision
  Other Names: AcuFocus Corneal Inlay ACI 7000 PDT; AcuFocus KAMRA inlay

SUMMARY:
The purpose of this study is to determine if the AcuFocus Corneal Inlay ACI 7000PDT will provide an effective method for the correction of presbyopia in patients who have normal distance vision but need a correction such as glasses or contact lenses to see clearly at near.

DETAILED DESCRIPTION:
The loss of near vision and the ability to perform tasks that require near vision is part of the normal aging process. This natural transformation in the eye occurs as a result of the loss of accommodation of the crystalline lens, a condition known as presbyopia. The crystalline lens is responsible for the accommodative properties of the human eye, as established by Young in 1801, over 200 years ago.1 During accommodation, the ciliary muscle contracts, decreasing tension on the zonules, and allowing the crystalline lens to thicken, increasing its refractive power. This mechanism of accommodation and thickening of the lens provides the eye with adequate refractive power for near vision. The loss of accommodation with aging is the result of changes in the crystalline lens composition that prevent the natural accommodative process from occurring. This is associated with the gradual loss of near vision without external correction, generally in the form of spectacles.

The AcuFocus™ ACI 7000PDT represents new technology based on the well-established concept of small-aperture optics. In early cameras, depth of focus was controlled by reducing the aperture through which light enters. The smaller the aperture, the greater the depth of focus will be. This concept also applies to the human eye. In the eye of a presbyopic emmetrope, the lens cannot accommodate sufficiently to focus the light rays from a near object onto a single point on the retina. Thus, a point object is imaged as a blur circle on the retina, and images of extended objects are degraded as well. If an opaque disc with a small aperture in the center is placed in front of the eye, the peripheral rays will be obscured while the central rays pass unaffected. Since peripheral rays enter the eye at a larger angle, they create a larger blur circle at the retinal image plane. Eliminating these peripheral rays reduces the size of the blur circle, improving image resolution.

In presbyopic subjects, objects closer than arm's length are focused behind the retina, thus creating blurred retinal images (which are composed of blur circles). A small aperture inlay placed in front of the eye of these subjects allows them to see at near by reducing the size of the blur circle.

AcuFocus, Inc. has developed a stationary intracorneal inlay designed to create a small aperture effect. The implant is intended to be placed intra-stromally either under a corneal flap or into a corneal pocket. Placement of the ACI will be centered over the pupil in the non-dominant eye. The ACI is expected to increase the depth of focus of the eye by reducing the circle of blur. Based on theoretical calculations of small aperture optics, the ACI is expected to provide presbyopic subjects with improvement of near and intermediate vision.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be natural emmetropes needing a minimum magnitude of +1.00D to +2.50D of reading add.
2. Subjects must have uncorrected near visual acuity worse than 20/40 and better than 20/100 in the eye to be implanted.
3. Subject must have distance visual acuity correctable to at least 20/20 in both eyes.
4. Subjects must have a preoperative spherical equivalent of plano defined as +0.50D to -0.75D with no more than 0.75D of refractive cylinder as determined by cycloplegic refraction in the eye to be implanted.

Exclusion Criteria:

1. Subjects with a difference of > 1.00D between the spherical equivalent manifest refraction and the spherical equivalent cycloplegic refraction.
2. Subjects with anterior segment pathology, including cataracts, in the eye to be implanted.
3. Subjects with residual, recurrent, active ocular or uncontrolled eyelid disease, or any corneal abnormalities (including endothelial dystrophy, guttata, recurrent corneal erosion, etc.) in the eye to be implanted.
4. Subjects with ophthalmoscopic signs of keratoconus (or keratoconus suspect) in the eye to be implanted.
5. Subjects with a history of chronic dry eye not responding to therapy.
6. Subjects with distorted or unclear corneal mires on topography maps of the eye to be implanted.
7. Subjects who require canthotomy to generate a corneal flap in the eye to be implanted.
8. Subjects with macular degeneration, retinal detachment, or any other fundus pathology that would prevent an acceptable visual outcome in the eye to be implanted.
9. Subjects who have undergone previous intraocular or corneal surgery including cataract and LASIK surgery.
10. Subjects with a history of herpes zoster or herpes simplex keratitis.
11. Subjects who have a history of steroid-responsive rise in intraocular pressure, preoperative IOP > 21 mmHg, glaucoma, or is a glaucoma suspect.
12. Subjects with a history of diagnosed diabetes, autoimmune disease, connective tissue disease, or clinically significant atopic syndrome.
13. Subjects on chronic systemic corticosteroids or other immunosuppressive therapy that may affect wound healing, and any immunocompromised subjects.
14. Subjects who are using ophthalmic medication(s) other than artificial tears for treatment of any ocular pathology including ocular allergy.
15. Subjects using systemic medications with significant ocular side effects.
16. Subjects who are pregnant, lactating, or of child-bearing potential and not practicing a medically approved method of birth control.
17. Subjects with known sensitivity to planned study concomitant medications.
18. Subjects who are participating in any other ophthalmic drug or device clinical trial during the time of this clinical investigation.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2009-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Perry Binder, MD, Study Director
Locations (8):
- Australia (2):
  - Vista Laser Eye Clinics, Melbourne, Victoria
  - The Eye Institute, Bondi Junction
- Paracelsus Medizinische Privat-Universität, PMU, Universitätsklinikum, Salzburg, Austria
- Universitats-Augenklinik, Department of Ophthalmology, Bochum, Germany
- New Zealand (2):
  - The Fendalton Eye Clinic, Fendalton, Christchurch
  - Auckland Eye, Auckland
- Singapore National Eye Centre, Singapore, Singapore
- Optical Express, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dexl AK, Seyeddain O, Riha W, Hohensinn M, Ruckl T, Hitzl W, Grabner G. Reading performance after implantation of a modified corneal inlay design for the surgical correction of presbyopia: 1-year follow-up. Am J Ophthalmol. 2012 May;153(5):994-1001.e2. doi: 10.1016/j.ajo.2011.08.044. Epub 2011 Nov 20. PMID 22105801
- See also: Sponsor website — http://www.acufocus.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 119 participants were consented for the study (enrolled), and 118 subsequently were implanted with the device (started) for the study.
Groups:
- AcuFocus Corneal Inlay: Implantation of the AcuFocus Corneal Inlay in emmetropic presbyopic patients.
  AcuFocus Corneal Inlay ACI 7000PDT: corneal inlay
Period: Overall Study
Arm/Group | AcuFocus Corneal Inlay
Started | 118
Completed | 101
Not Completed | 17

BASELINE CHARACTERISTICS:
Population: Patients between 45 and 60 years of age with presbyopia
Groups:
- AcuFocus Corneal Inlay: Implantation of the AcuFocus Corneal Inlay in emmetropic presbyopic patients.
  AcuFocus Corneal Inlay ACI 7000PDT: Inlay implanted in cornea for improvement of near vision
Arm/Group | AcuFocus Corneal Inlay
Number analyzed (Participants) | 118
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 118
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 67
Region of Enrollment [Count of Participants; unit: Participants]
  New Zealand | 18
  Austria | 24
  Singapore | 9
  United Kingdom | 11
  Australia | 42
  Germany | 3
  Philippines | 11

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Uncorrected Near Visual Acuity
Description: Percent of subjects who achieved UCNVA of 20/40 or better.
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | AcuFocus Corneal Inlay
Number analyzed (Participants) | 118
percentage of participants | 78.2

2. Secondary Outcome: Improvement of Near Uncorrected Visual Acuity
Description: Mean subjective rating via questionnaire on 1 to 7 rating scale (1= very dissatisfied and 7 = very satisfied).
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AcuFocus Corneal Inlay
Number analyzed (Participants) | 118
units on a scale | 4.7 (1.7)

ADVERSE EVENTS:
Time Frame: 3 months, 6 months, 1 year, 2 years,3 years
Arm/Group | AcuFocus Corneal Inlay
Serious Adverse Events (participants affected / at risk) | 4/118
Other Adverse Events (participants affected / at risk) | 52/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AcuFocus Corneal Inlay (N=118)
Hospitalization secondary to prostatectomy (Surgical and medical procedures) | 1 (1)
Hospitalization due to bike accident (Injury, poisoning and procedural complications) | 1 (1)
Stromal thinning secondary to abnormal healing response to corneal trauma (Eye disorders) | 1 (1)
Hip replacement surgery (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AcuFocus Corneal Inlay (N=118)
Blepharitis (Infections and infestations) | 1 (1)
Superficial punctate keratitis (Eye disorders) | 2 (2)
Flap complication (Surgical and medical procedures) | 2 (2)
Vision (Eye disorders) | 9 (9) — Decrease in BCDVA greater than 2 lines month 3 and later
Cornea (Eye disorders) | 8 (8) — Corneal edema
Secondary Surgical Intervention (Surgical and medical procedures) | 2 (2) — Inlay recentration
Secondary Surgical Intervention (Surgical and medical procedures) | 1 (1) — Epithelial ingrowth removal
Intraocular Pressure (Eye disorders) | 5 (5)
Conjunctivitis (Eye disorders) | 2 (2)
Hordeolum (Eye disorders) | 1 (1)
Limbal foreign body (Eye disorders) | 1 (1)
Corneal abrasion/erosion (Eye disorders) | 1 (1)
Foreign bodies over inlay with anterior corneal surface defect (Eye disorders) | 1 (1)
Lens (Eye disorders) | 1 (1) — Cataract
Meibomian Gland Dysfunction (Eye disorders) | 1 (1)
Partial sidecut at inner edge of mask (Eye disorders) | 1 (1)
Admission to hospital for severe headache (General disorders) | 1 (1)
Hypercholesterolemia (General disorders) | 1 (1)
Increased blood sugar (General disorders) | 1 (1)
Hypertension (General disorders) | 2 (2)
Scleroderma (General disorders) | 1 (1)
Chest Infection (General disorders) | 1 (1)
Knee injury & surgery (Surgical and medical procedures) | 1 (1)
Non-insulin-dependent diabetes mellitus (General disorders) | 1 (1)
Benign Prostate Hyperplasia (General disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1) — Fellow eye
Conjunctival Cyst (Eye disorders) | 1 (1) — Fellow Eye
Upper eyelid chalazion (Eye disorders) | 1 (1) — Fellow eye

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other